CLINICAL TRIAL: NCT02796105
Title: Evaluation of Efficacy and Safety of Medroxiprogesterone Acetate (Progevera 10 mg®) Versus GnRh Antagonist (Orgalutran®) in Ovarian Stimulation Cycles of Oocyte Donors
Brief Title: Progevera 10 mg® Versus Orgalutran® in Ovarian Stimulation Cycles of Oocyte Donors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Privada Eugin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRAKE
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — ganirelix

ARMS (2):
- Progevera (Experimental): Progevera 10 mg
  Interventions: Drug: Progevera
- Orgalutran (Active Comparator): Orgalutran 0.25 mg
  Interventions: Drug: Orgalutran

INTERVENTIONS:
Drug: Progevera
  Arms: Progevera
Drug: Orgalutran
  Arms: Orgalutran

SUMMARY:
Evaluation of efficacy and safety of medroxiprogesterone acetate (Progevera 10 mg®) versus GnRh antagonist (Orgalutran®) in ovarian stimulation cycles of oocyte donors

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors included in the oocyte donation program of Clinica EUGIN.
* 1st oocyte donation cycle at Clínica EUGIN.

Exclusion Criteria:

* Polycistic Ovarian syndrome (PCOs).
* Estradiol levels on day 2 of menstrual cycle >70 pg/ml.
* Hormone treatments up to 3 months before the oocyte donation cycle.
* Medical contraindication to the treatments used in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
donor ovarian response | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca Begueria, Dr, Principal Investigator — Clinica Eugin
Locations (1):
- Clinica Eugin, Barcelona, Spain

REFERENCES:
- [Derived] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417